CLINICAL TRIAL: NCT03067454
Title: Early Mobilization of Spiral Metacarpal Fractures Compared With Operative Treatment - a Prospective Randomized Trial
Brief Title: Early Mobilization of Spiral Metacarpal Fractures Compared With Operative Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FOU 2017-0056
Record Dates: First submitted 2017-02-21; First posted 2017-03-01 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Fracture
Keywords: early mobilisation; metacarpal fracture; operation
MeSH Terms: conditions — Fractures, Bone | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Prospective randomised controlled trial to compare operation and treatment with early mobilisation for metacarpalfractures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conservative group (Other): Treatment with early mobilisation
  Interventions: Procedure: Early mobilisation
- operative group (Other): Treatment with operation
  Interventions: Procedure: Operation

INTERVENTIONS:
Procedure: Early mobilisation — Conservative treatment with early mobilisation
  The patient is instructed to do a fist and is not allowed to leave the clinic before. Active mobilisation under control (doctor or physiotherapist) is performed until healing of the fracture is documented.
  Arms: conservative group
Procedure: Operation — Operation of the fracture. Usually open reduction and internal fixation with plates and screws or just screws within 2 weeks of injury. Immobilisation in a cast for two weeks followed by physiotherapy.
  Arms: operative group

SUMMARY:
Spiral metacarpal fractures (metacarpal II-V) can be treated conservatively or with operation. With minimal displacement this fracture is usually treated with immobilisation or early mobilisation. With appreciable displacement especially any malrotation the patient usually is treated with an operation. This usually includes an open reduction of the fracture and fixation with plates and screws or just screws. Even if this is an standard procedure both mild and severe complications have been reported. New studies have shown that even displaced fractures can be treated with early mobilization. In those cases the fractures may heal with some shortening but very good function. An advantage of early mobilization is that the patient avoids the risk of an operation and the costs for the treatment are decreased markedly. The study is designed to answer the question if early mobilization is not inferior to operative treatment but with lower costs and without any operation related risks.

DETAILED DESCRIPTION:
The study is designed as an prospective, randomised controlled trial. The patients are divided into two groups (operative and conservative treatment with early mobilisation). The operative group is treated with internal fixation and 2 weeks in a cast. The conservative group is instructed to do a fist to correct any malrotation and to rehabilitate quickly. By this procedure shortening oft he metacarpalfractures is limited by the function of the deep transverse metacarpal ligament connecting the distal parts of the metacarpalbones II-V. Furthermore the participants in the conservative group are allowed to use their hands without any restrictions. A physiotherapist controls that early mobilisation is carried out.

The participant will be seen for a follow-up at 1, 6 and 12 weeks and 1 year. Radiographs will be performed at 1v and 6v. The finger ranges of motion and pain will be evaluated with every follow-up, DASH score, range of motion, pain and grip-strength will be measured after 12v and 1 year. The investigators will measure return to driving, work and sport.

Complications will be registered continuously for all patients. The overall satisfaction of the patients and the costs for both treatments will be documented as well.

The study population is planned to be 21 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

* single spiral fractures of metacarpal bone II-V
* fracture line at least twice the length of the diameter of the bone at the level of the fracture
* at least 1-2mm displacement of the fracture and/or malrotation
* normal hand function before the injury
* fracture less than 10 days old

Exclusion Criteria:

* multiple metacarpal fractures
* open fractures
* incompliance or dementia
* fracture line not twice the length of the diameter of the bone at the level of the fracture
* abnormal hand function before the injury
* fracture more than 10 days old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Grip-strength measured by the JAMAR dynamometer | 1 year
  Power of the treated hand measured by the JAMAR dynamometer compared with the none-operated hand

SECONDARY OUTCOMES:
Handfunction rated by the DASH-score | 1 year
  DASH-score
Range of motion in the treated hand/fingerray | 1 year
  Range of motion in the treated hand measured in degrees of active motion with a hand held goniometer (operated fingerray)
Appearance and severity of complications | 1 year
  Complications during the different treatments
Time until the patient can return to work, driving and sport | 1 year
  Return to work, driving and sport
The total costs of each treatment | 1 year
  Costs of each treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nils Hailer, Professor, Study Director — Department of Orthopedics, Uppsala University Hospital; Daniel Muder, MD, Dr. med., Principal Investigator — Department of Orthopedics, Falu lasarett; Grey Giddins, M.B.B.Ch. F.R.C.S. (Orth), Principal Investigator — Royal United Hospitals Bath NHS Foundation Trust
Locations (2):
- Sweden (2):
  - Falu lasarett, Department of Orthopedics, Falun, Dalarna County
  - Uppsala University Hospital, Dept. of Handsurgery, Uppsala, Uppsala County

IPD SHARING:
Plan to Share IPD: No